CLINICAL TRIAL: NCT02394158
Title: Preventing Recurrent Gestational Diabetes Mellitus With Early Metformin Intervention
Brief Title: Preventing Recurrent Gestational Diabetes With Metformin
Acronym: PRoDroME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); London North West Healthcare NHS Trust (Other); The Novo Nordisk UK Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14SM1971; 2014-001244-38 (EudraCT Number)
Record Dates: First submitted 2015-03-02; First posted 2015-03-20 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Recurrent Gestational Diabetes Mellitus; Prevention; Metformin
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm Metformin (Active Comparator): Metformin (500mg tablets) to start at a dose of 500mg once daily with an increase of 500mg every five days until the maximum dose of 1000mg twice daily is reached.
  Interventions: Drug: Metformin
- Control arm placebo (Placebo Comparator): Matched placebo tablets (500mg) to start at a dose of 500mg once daily with an increase of 500mg every five days until the maximum dose of 1000mg twice daily is reached.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metformin
  Arms: Intervention arm Metformin
Drug: placebo
  Arms: Control arm placebo

SUMMARY:
Study Hypothesis: Intervention with metformin therapy early in pregnancy will prevent gestational diabetes mellitus recurring in previously affected pregnancies.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is a common medical complication of pregnancy and is associated with increased risks to mother and baby. The incidence is increasing reflecting changing pre-gravid female demographics. Once one pregnancy is complicated by GDM, subsequent pregnancies are more likely to be affected by the same condition. This reported risk of recurrence is estimated to range between 35 and 80%, with non-caucasian ethnicity being the strongest predictor of GDM recurrence. Evidence regarding further predictors of recurrent GDM is conflicting and measures that might prevent recurrence need exploring.

Metformin is commonly used in the treatment of established GDM and has been shown to reduce the incidence of GDM in the context of polycystic ovarian syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy;
* 8-22 weeks gestation
* Previous pregnancy complicated by gestational diabetes

Exclusion Criteria:

* Established pre-existing diabetes (including unrecognised diabetes defined as a fasting plasma glucose ≥ 7.0mmol/L and/ or HbA1c ≥ 48mmol/mol); Contraindications to metformin therapy (creatinine ≥ 130μmol/L/ alanine transaminase ≥ 2.0 x upper limit normal/ previous intolerance to metformin)
* Planned continued antenatal care/ delivery at centre not included in trial
* Planned fast for cultural/ religious reasons e.g. Ramadan

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Singleton pregnancy; in 8-22 weeks gestation, previous pregnancy complicated by gestational diabetes
Enrollment: 112 (Estimated)
Dates: Start 2015-01-27 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Development of Gestational Diabetes at any point during the course of pregnancy | From 12 weeks pregnancy until the onset of labour

SECONDARY OUTCOMES:
Maternal gestational weight gain | Difference between weight at 12 weeks gestation and 36 weeks gestation
Requirement for insulin therapy | From 12 weeks gestation until 36 weeks gestation
Postpartum glucose levels | 6 weeks postpartum
Levels of maternal physical and psychological health as assessed by questionnaires | From 12 weeks gestation until 6 weeks postpartum
Fetal birthweight and birthweight centile | At Birth
Composite of neonatal outcomes (neonatal hypoglycaemia requiring treatment, respiratory distress syndrome requiring oxygen therapy/ continuous positive airway pressure, neonatal hyperbilirubinaemia requiring phototherapy). | At Birth
Cost effectiveness of the intervention | From 12 weeks gestation until 6 weeks postpartum
  Difference in requirement for medical services and unplanned hospital/ General Practitioner attendances between the two arms

OTHER OUTCOMES:
Insulin resistance | From 12 weeks gestation until 6 weeks postpartum
Maternal triglyceride concentrations | From 12 weeks gestation until 6 weeks postpartum
Fetal hyperinsulinaemia | Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Robinson, FRCP, MD, Principal Investigator — Imperial College NHS Trust
Locations (2):
- United Kingdom (2):
  - Imperial College NHS Trust, London
  - London North West Healthcare Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Rowan JA, Hague WM, Gao W, Battin MR, Moore MP; MiG Trial Investigators. Metformin versus insulin for the treatment of gestational diabetes. N Engl J Med. 2008 May 8;358(19):2003-15. doi: 10.1056/NEJMoa0707193. PMID 18463376
- [Background] Getahun D, Fassett MJ, Jacobsen SJ. Gestational diabetes: risk of recurrence in subsequent pregnancies. Am J Obstet Gynecol. 2010 Nov;203(5):467.e1-6. doi: 10.1016/j.ajog.2010.05.032. Epub 2010 Jul 13. PMID 20630491
- [Background] Thangaratinam S, Rogozinska E, Jolly K, Glinkowski S, Roseboom T, Tomlinson JW, Kunz R, Mol BW, Coomarasamy A, Khan KS. Effects of interventions in pregnancy on maternal weight and obstetric outcomes: meta-analysis of randomised evidence. BMJ. 2012 May 16;344:e2088. doi: 10.1136/bmj.e2088. PMID 22596383
- [Background] De Leo V, Musacchio MC, Piomboni P, Di Sabatino A, Morgante G. The administration of metformin during pregnancy reduces polycystic ovary syndrome related gestational complications. Eur J Obstet Gynecol Reprod Biol. 2011 Jul;157(1):63-6. doi: 10.1016/j.ejogrb.2011.03.024. Epub 2011 May 6. PMID 21530058